CLINICAL TRIAL: NCT05726942
Title: Efficacy of mHealth Applications in Weight Management in a Population Affected by Overweight or Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HS-2022-0256
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Overweight and Obesity
Keywords: adiposity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthi (Experimental)
  Interventions: Other: Healthi
- Control (No Intervention)

INTERVENTIONS:
Other: Healthi — Healthi refers to the Healthi app, which is a mobile application for weight loss
  Arms: Healthi

SUMMARY:
The purpose of this study is to determine the effectiveness of mobile health applications in improving health outcomes in patients with overweight and obesity. This study will involve a 6-month long commitment where participants will be expected to use an mHealth app daily, weigh themselves and check their fasting blood glucose levels every morning.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18-64
* BMI ≥ 25
* Owns or has access to a bathroom weight scale
* Owns a smartphone and willing to download mobile app

Exclusion Criteria:

* On medications that promote weight gain such as antipsychotic, antidepressant, and steroid hormone medications.
* Medications for diabetes such as insulin, thiazolidinediones or sulfonylureas are okay

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of mHealth apps at changing bodyweight assessed by bodyweight measurements over 6 months | 3 months
  Determine if the mhealth app is an effective weight loss modality compared to standard weight loss program (control)
  Outcome measure will be body weight in kg
Self-efficacy in weight management assessed by Weight Management and Nutrition Knowledge questionnaire | 3 months
  Compare and determine which intervention promotes self-efficacy in weight management.
  Reporting will be on a scale of 0-100, with higher scores indicating higher self-efficacy
Long-term change in diabetes via fasting blood glucose | 3 months
  Compare and determine which intervention elicits the most change towards diabetes via fasting blood glucose
  Outcome measure will be fasting blood glucose
Quality of Life after using mHealth apps assessed by World Health Organization Quality of Life BREF questionnaire | 3 months
  Comparing the two arms to determine which leads to greater quality of life (QOL)
  Measures will be reported on a scale of 1-5 across four domains. Scores will be converted to a scale of 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No